CLINICAL TRIAL: NCT03695198
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3361237 in Healthy Subjects
Brief Title: A Study of LY3361237 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16969; I9S-MC-BTAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3361237 - Subcutaneous (SC) (Experimental): LY3361237 administered SC
  Interventions: Drug: LY3361237 - SC
- Placebo - SC (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo - SC
- LY3361237 - Intravenous (IV) (Experimental): LY3361237 administered IV
  Interventions: Drug: LY3361237 - IV
- Placebo - IV (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo - IV

INTERVENTIONS:
Drug: LY3361237 - SC — LY3361237 administered SC
  Arms: LY3361237 - Subcutaneous (SC)
Drug: LY3361237 - IV — LY3361237 administered IV
  Arms: LY3361237 - Intravenous (IV)
Drug: Placebo - SC — Placebo administered SC
  Arms: Placebo - SC
Drug: Placebo - IV — Placebo administered IV
  Arms: Placebo - IV

SUMMARY:
The purposes of this study are to determine:

* The safety of LY3361237 and any side effects that might be associated with it.
* How much LY3361237 gets into the blood stream and how long it takes the body to remove it in healthy participants.

Participants will be admitted to the clinical research unit (CRU) for 4 overnight stays. The study will last about 12 weeks for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, as determined by medical history and physical examination.
* To qualify as Japanese for this study, the participant, the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan.
* Between 18 (20 for Japanese participants) and 65 years of age.
* Have a body mass index of 18.0 to 32.0 kilograms per meter squared, inclusive, and a minimum body weight of 45.0 kilograms.

Exclusion Criteria:

* Show evidence of active or latent tuberculosis (TB), as documented by medical history and examination, chest x-ray and TB testing
* Are immunocompromised
* Have evidence of chronic viral infection have received live vaccine(s) (including attenuated live vaccines) within 28 days of screening or intend to receive during the study (non-live or inactivated vaccinations are allowed). Bacillus Calmette-Guérin (BCG) vaccine must not have been administered within 12 months of screening
* Have had lymphoma, leukemia, or any malignancy or pre-malignant condition within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 12
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3361237 | Predose through Week 12
  PK: Cmax of LY3361237
PK: Area Under the Plasma Concentration Time Curve (AUC) of LY3361237 | Predose through Week 12
  PK: AUC of LY3361237

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No